CLINICAL TRIAL: NCT01216670
Title: Cardiac Rhythm Monitoring After Acute Decompensation for Heart Failure
Acronym: CARRYINGON
Status: Completed | Type: Observational
Sponsor: Medtronic Italia (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT-CARRYINGONforHF
Record Dates: First submitted 2010-04-21; First posted 2010-10-07 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2013-02

CONDITIONS: Heart Failure
Keywords: Reveal® XT; Acute Heart Failure; Low Ejection Fraction; Reveal® XT implanted
MeSH Terms: conditions — Heart Failure | interventions — Blood Glucose Self-Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: remote patient's management — scheduled remote CareLink data transmission
  Other Names: home monitoring

SUMMARY:
The CARRYING ON for heart failure (HF) study is a national, prospective, post market interventional, multi-center, open-label, pilot trial.The purpose of the study is to assess a short term and a long term period, incidence of pre-specified clinical and arrhythmic events in patients with a low ejection fraction (EF) that are hospitalized for acute cardiac decompensation.

DETAILED DESCRIPTION:
The CARRYING ON for heart failure (HF) study is a national, prospective, post market interventional, multi-center, open-label, pilot trial designed in two phases.

The purpose of the study is to assess a short term (6 months follow-up - Phase 1) and a long term period (24 months follow-up - Phase 2), incidence of pre-specified clinical and arrhythmic events in patients with a low ejection fraction (EF) that are hospitalized for acute cardiac decompensation. A previously implanted Reveal® XT device will be used to collect heart rhythm information.

ELIGIBILITY:
Inclusion Criteria:

* Subject with a history of at least one heart failure (HF) hospitalization (as defined in the European Society of Cardiology or American College of Cardiology/American Heart Association guidelines), emergency department (ED) visit, or urgent office visit necessitating intravenous (IV) diuretic or augmentation of oral diuretic, IV inotropic, or IV vasodilator or other HF parenteral therapy within 15 days prior to device implant
* Subject has an implanted Reveal® XT device (less than 15 days post implant);
* Ejection Fraction (EF) less than 40 percent
* Patient with access to a telephone line
* Patient or the patient's caregiver is willing and able to use the Medtronic CareLink® Network Monitor and to perform the required duties at home or has a family member or assistant perform those duties
* Age greater than 18 years old
* Patient is willing and able to comply with the Clinical Investigation plan and willing to remain available for follow-up visit, through study closure
* Patient (or patient's legally authorized representative) is willing and able to sign and date the study Informed Consent

Exclusion Criteria:

* New York Heart Association (NYHA) Class IV (chronic or ambulatory)
* Planned or previous implant of implantable cardioverter-defibrillator or pacemaker device
* Patient's life expectancy is less than one year due to non cardiovascular disorders, in the opinion of the physician
* Severe chronic obstructive pulmonary disorder (COPD)
* Chronic Atrial Fibrillation at time of enrollment
* ST segment elevation at time of electrocardiogram
* Cognitive disease
* Pregnancy or childbearing potential and not on reliable contraceptive
* Anticipated compliance problem or participation in another competitive trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hf patients without indication to permanent device implant (PM/ICD/CRT)
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2011-02; Primary Completion 2013-11 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Phase I: incidence of pre-specified clinical and arrhythmic events | implant to 6 months post-implant
  In patients with low ejection fraction that are hospitalized for acute cardiac decompensation, the pre-specified events include:
  1. Cardiovascular mortality or unplanned cardiovascular hospitalizations (including hospitalizations that will be scheduled due to pacemaker, implantable cardioverter-defibrillator, or cardiac resynchronization therapy device implant)
  2. Arrhythmic events
Phase II: incidence of pre-specified clinical and arrhythmic events | implant to 24 months post-implant
  In patients with low ejection fraction that are hospitalized for acute cardiac decompensation, the pre-specified events include:
  1. Cardiovascular mortality or unplanned cardiovascular hospitalizations (including hospitalizations that will be scheduled due to pacemaker, implantable cardioverter-defibrillator, or cardiac resynchronization therapy device implant)
  2. Arrhythmic events

SECONDARY OUTCOMES:
Phase I: incidence of the pre-specified secondary clinical and arrhythmic events in patients implanted with the Reveal® XT | implant to 6 months post-implant
  Document the incidence of the pre-specified secondary clinical and arrhythmic events in patients implanted with the Reveal XT.
  The pre-specified secondary clinical and arrhythmic events are:
  * Time to first detection of brady-tachyarrhythmia episode;
  * All cause mortality or unplanned cardiovascular hospitalization;
  * Unplanned cardiovascular hospitalization;
  * Heart Failure hospitalization;
  * Cardiovascular mortality;
  * Serious cardiovascular Adverse Events.
Phase II: incidence of the pre-specified secondary clinical and arrhythmic events in patients implanted with the Reveal® XT | implant to 24 months post-implant
  Document the incidence of the pre-specified secondary clinical and arrhythmic events in patients implanted with the Reveal XT.
  The pre-specified secondary clinical and arrhythmic events are:
  * Time to first detection of brady-tachyarrhythmia episode;
  * All cause mortality or unplanned cardiovascular hospitalization;
  * Unplanned cardiovascular hospitalization;
  * Heart Failure hospitalization;
  * Cardiovascular mortality;
  * Serious cardiovascular Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: CARRYING ON Study Trial Leader, Study Chair — Medtronic
Locations (4):
- Italy (4):
  - A.O. SS. Antonio e Biagio e Cesare Arrigo di Alessandria, Alessandria, Alessandria
  - A.O. Ospedale S. Anna di Como, Como, Como
  - Policlinico di Monza, Monza, Monza
  - Clinica San Gaudenzio, Novara, Novara

REFERENCES:
- [Background] Fonarow GC; ADHERE Scientific Advisory Committee. The Acute Decompensated Heart Failure National Registry (ADHERE): opportunities to improve care of patients hospitalized with acute decompensated heart failure. Rev Cardiovasc Med. 2003;4 Suppl 7:S21-30. PMID 14668697
- [Background] Nieminen MS, Bohm M, Cowie MR, Drexler H, Filippatos GS, Jondeau G, Hasin Y, Lopez-Sendon J, Mebazaa A, Metra M, Rhodes A, Swedberg K, Priori SG, Garcia MA, Blanc JJ, Budaj A, Cowie MR, Dean V, Deckers J, Burgos EF, Lekakis J, Lindahl B, Mazzotta G, Morais J, Oto A, Smiseth OA, Garcia MA, Dickstein K, Albuquerque A, Conthe P, Crespo-Leiro M, Ferrari R, Follath F, Gavazzi A, Janssens U, Komajda M, Morais J, Moreno R, Singer M, Singh S, Tendera M, Thygesen K; ESC Committe for Practice Guideline (CPG). Executive summary of the guidelines on the diagnosis and treatment of acute heart failure: the Task Force on Acute Heart Failure of the European Society of Cardiology. Eur Heart J. 2005 Feb;26(4):384-416. doi: 10.1093/eurheartj/ehi044. Epub 2005 Jan 28. No abstract available. PMID 15681577
- [Background] Di Lenarda A, Scherillo M, Maggioni AP, Acquarone N, Ambrosio GB, Annicchiarico M, Bellis P, Bellotti P, De Maria R, Lavecchia R, Lucci D, Mathieu G, Opasich C, Porcu M, Tavazzi L, Cafiero M; TEMISTOCLE Investigators. Current presentation and management of heart failure in cardiology and internal medicine hospital units: a tale of two worlds--the TEMISTOCLE study. Am Heart J. 2003 Oct;146(4):E12. doi: 10.1016/S0002-8703(03)00315-6. PMID 14564335
- [Background] Tavazzi L, Maggioni AP, Lucci D, Cacciatore G, Ansalone G, Oliva F, Porcu M; Italian survey on Acute Heart Failure Investigators. Nationwide survey on acute heart failure in cardiology ward services in Italy. Eur Heart J. 2006 May;27(10):1207-15. doi: 10.1093/eurheartj/ehi845. Epub 2006 Apr 7. PMID 16603579
- [Background] O'Connor CM, Stough WG, Gallup DS, Hasselblad V, Gheorghiade M. Demographics, clinical characteristics, and outcomes of patients hospitalized for decompensated heart failure: observations from the IMPACT-HF registry. J Card Fail. 2005 Apr;11(3):200-5. doi: 10.1016/j.cardfail.2004.08.160. PMID 15812748
- [Background] Cleland JG, Swedberg K, Follath F, Komajda M, Cohen-Solal A, Aguilar JC, Dietz R, Gavazzi A, Hobbs R, Korewicki J, Madeira HC, Moiseyev VS, Preda I, van Gilst WH, Widimsky J, Freemantle N, Eastaugh J, Mason J; Study Group on Diagnosis of the Working Group on Heart Failure of the European Society of Cardiology. The EuroHeart Failure survey programme-- a survey on the quality of care among patients with heart failure in Europe. Part 1: patient characteristics and diagnosis. Eur Heart J. 2003 Mar;24(5):442-63. doi: 10.1016/s0195-668x(02)00823-0. PMID 12633546
- [Background] Fonarow GC, Stough WG, Abraham WT, Albert NM, Gheorghiade M, Greenberg BH, O'Connor CM, Sun JL, Yancy CW, Young JB; OPTIMIZE-HF Investigators and Hospitals. Characteristics, treatments, and outcomes of patients with preserved systolic function hospitalized for heart failure: a report from the OPTIMIZE-HF Registry. J Am Coll Cardiol. 2007 Aug 21;50(8):768-77. doi: 10.1016/j.jacc.2007.04.064. Epub 2007 Aug 6. PMID 17707182
- [Background] Braunschweig F. Therapeutic and diagnostic role of electrical devices in acute heart failure. Heart Fail Rev. 2007 Jun;12(2):157-66. doi: 10.1007/s10741-007-9019-0. PMID 17447136
- [Derived] Vanoli E, Mortara A, Diotallevi P, Gallone G, Mariconti B, Gronda E, Gentili A, Bisetti S, Botto GL. Cardiac Rhythm Monitoring After Acute Decompensation for Heart Failure: Results from the CARRYING ON for HF Pilot Study. JMIR Res Protoc. 2016 Apr 26;5(2):e62. doi: 10.2196/resprot.4380. PMID 27118481